CLINICAL TRIAL: NCT00700414
Title: International Pediatric Adrenocortical Tumor Registry
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IPACTR
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Adrenocortical Tumor
MeSH Terms: conditions — Adrenal Cortex Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample with DNA and RNA; Tumor Tissue (of any histology); Adrenocortical tumors;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Any participant who meets eligibility criteria and consents to participate in the trial.

SUMMARY:
This study aims to collect demographic and medical information including detailed family history of cancer of children and adolescents with adrenocortical tumors in order to learn more about the clinical and epidemiological aspects, treatment modalities, and outcome of patients with this rare disease, worldwide.

In addition, investigators at St. Jude Children's Research Hospital (SJCRH) plan to perform molecular studies of tumor cells aimed to clarify the role of the TP53 gene and other genetic pathways in these tumors. They aim to obtain relevant biological material from participants with adrenocortical tumor (ACT), their biological parents, and relatives for determination of the TP53 germline status, molecular studies of the TP53 gene, and other molecular pathways.

DETAILED DESCRIPTION:
Adrenocortical tumors (ACT) are rare cancer types that form in the outer layer of the adrenal gland and are very uncommon in children and teenagers. There is variation in pediatric ACT incidence worldwide. In the United States, only about 25 new cases of ACT per million per year, making this a very rare tumor. However, in southern Brazil, the annual incidence of ACT is 15 times that seen in the United States accounting for 3.4-4.2 per million per year.

Molecular studies have revealed that the majority of children with ACT, particularly those younger than 4 years of age, have constitutional TP53 mutations and/or imprinting defects at chromosome 11p as observed in Beckwith Wiedemann syndrome (BWS) patients. Some mutations, as exemplified by the R337H TP53 germline mutation, in which the function of the mutant protein is relatively preserved, the history of cancer in the carriers and their families is relatively unremarkable. In other cases, the TP53 mutated gene encodes a functionally-impaired protein that predicts for a pervasive history of familial cancer (Li-Fraumeni syndrome). Therefore, these observations have implications for genetic counseling of families with childhood ACT and underscore the importance of genotype-phenotype correlations in familial cancer syndromes.

The creation of a rare tumor registry provides a mechanism to collect information that cannot be gathered in a single institution. The analysis of the registry data would permit an overview of the clinical, epidemiological, current treatment standards, and survival data of these patients and thus create opportunities for research. It also may facilitate the development of treatment consensus among investigators who register their patients and help to design future studies. Moreover, the combined Children's Oncology Group (COG) and IPACTR studies are expected to provide meaningful insight into the biology of ACT, including clinical phenotype/genotype relationships, treatment outcome and long-term follow-up data in subjects with this rare tumor. Finally, it would provide data on the long-term consequences of exposure to tumor-secreted androgens (found in more than 80% of the pediatric cases) on children's growth and development.

ELIGIBILITY:
STRATIFICATION ASSIGNMENT:

* Stratum A: participant suspected or confirmed diagnosis of adrenocortical tumor (ACT)
* Stratum R: relative of participant with ACT and TP53 mutation who has diagnosis of malignancy
* Stratum P: biological parent of participant with ACT

Inclusion Criteria - Stratum A (participant with ACT):

* Age ≤ 21 years old at diagnosis
* Suspected or confirmed diagnosis of adrenocortical tumor (adenoma, carcinoma or undefined histology).
* Signed informed consent

Inclusion Criteria - Stratum R (relative):

* Any age
* Diagnosis of malignant tumor
* Signed informed consent

Inclusion Criteria - Stratum P (parent):

* Biological parent of Stratum A participant

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Age ≤ 21 years old at diagnosis of adrenocortical tumor.
  Relatives of the ACT patients of any age with a diagnosis of malignant tumor.
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 2001-10-01 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Collect demographic/medical information, detailed family history of cancer of children/adolescents with adrenocortical tumors, learn more about the clinical and epidemiological aspects, treatment modalities, and outcome of patients | Annually from diagnosis until no longer being followed, defined as up to 5 years from the date of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Raul C Ribeiro, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - All Children's Hospital/St. Petersburg Hospital, St. Petersburg, Florida
  - The Children's Medical Center, Dayton, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

REFERENCES:
- [Derived] Pinto EM, Maxwell KN, Halalsheh H, Phillips A, Powers J, MacFarland S, Walsh MF, Breen K, Formiga MN, Kriwacki R, Nichols KE, Mostafavi R, Wang J, Clay MR, Rodriguez-Galindo C, Ribeiro RC, Zambetti GP. Clinical and Functional Significance of TP53 Exon 4-Intron 4 Splice Junction Variants. Mol Cancer Res. 2022 Feb;20(2):207-216. doi: 10.1158/1541-7786.MCR-21-0583. Epub 2021 Oct 21. PMID 34675114
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols